CLINICAL TRIAL: NCT06118567
Title: Nitrous Oxide and Cortico-Limbic Function in Aggression
Brief Title: Effect of Nitrous Oxide on Aggression.
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Ohio State University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Emil Coccaro, Professor, Ohio State University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 2020H0368
Record Dates: First submitted 2023-11-01; First posted 2023-11-07 (Actual); Last update posted 2025-03-27 (Actual); Status verified 2025-03

CONDITIONS: Intermittent Explosive Disorder
Keywords: IED
MeSH Terms: conditions — Disruptive, Impulse Control, and Conduct Disorders | interventions — Nitrous Oxide

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Room air (vs. Nitrous Oxide Inhalation)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Nitrous Oxide Inhalation (Active Comparator): 60 minute session inhaling Nitrous Oxide gas.
  Interventions: Drug: Nitrous oxide
- Room Air (Sham Comparator): 60 minute session inhaling Room Air.
  Interventions: Drug: Room Air

INTERVENTIONS:
Drug: Nitrous oxide — Nitrous oxide gas.
  Arms: Nitrous Oxide Inhalation
Drug: Room Air — Room Air
  Arms: Room Air

SUMMARY:
The goal of this experimental medicine clinical trial is to test the hypothesis that nitrous oxide inhalation will result in a change in neurocircuit function in healthy controls and in individuals with impulsive aggressive tendencies. The main question aims to answer are: Does Nitrous Oxide normalize brain circuit function in impulsively aggressive individuals 24 hours after inhalation. Participants will undergo a 60 minute inhalation session with 50% Nitrous Oxide (or room air at another session) and then undergo an fMRI scan 24 hours later. Researchers will compare healthy controls and impulsively aggressive individuals to see if Nitrous Oxide can normalize the function of cortico-limbic circuits in the latter group.

DETAILED DESCRIPTION:
This study is designed to see if inhalation of 50% nitrous oxide (N2O) also known as laughing gas, can normalize cortico-limbic circuit functioning in impulsively aggressive human subjects. If the study results are positive, it would allow further studies of this potential treatment modality for those with recurrent, problematic, impulsive aggressive behavior (Intermittent Explosive Disorder: IED). IED is a disorder in which there are frequent and sudden outbursts of anger (yelling, throwing and breaking things, hitting people) that lead to problems with other people socially or at work. It affects about 4% of the US population lifetime, and does not have any approved treatments. The study will test if N2O can normalize brain activity 24 hours after infusion, in participants with a diagnosis of IED compared with healthy, non-aggressive, controls. This is a double-blinded-randomized study with comparison between groups (controls and IED patients) and comparison for each participant between N2O and placebo (air) inhalation. Participants will receive one type of inhalation 24 hours before undergoing an fMRI. Participants will be randomized to the order in which they receive N2O or air. Participants and study personnel involved in collection of outcome measures will be blinded to the type of inhalation. The study includes up to 7 visits. Visits 1/2 include interviews and questionnaires. At visits 3 and 5, participants receive the N2O or air inhalation. At visits 4 and 6, participants undergo fMRI while completing computer tasks. Visit 7 is to assure data collection is complete.

ELIGIBILITY:
Inclusion Criteria:

All participants:

* Between 21 and 55 years of age.
* Physically healthy (no clinically significant medical condition as confirmed by medical history/physical exam).
* Able to give informed consent.

Aggressive (IED) Study Participants (n = 25 Completed; 75 Enrolled).

* Current DSM-5 Criteria for IED
* LHA Aggression scores > 12
* Negative for a history of psychosis, bipolar disorder, developmental disorder, intellectual disability or a current substance use disorder.

Healthy, Non-Aggressive, Controls (n = 25 Completed, 75 Enrolled).

* Do not meet current/lifetime DSM-5 Criteria for any psychiatric disorder
* LHA aggression scores < 12

Exclusion Criteria:

* PCL Screening Version Score > 13; i.e., subject is likely to be psychopathic.32
* Current DSM-5 Major Depressive Episode.
* Life history of bipolar disorder/schizophrenia/organic mental syndrome.
* Intellectual disability [i.e., IQ < 70].
* History of N2O abuse/dependence.
* Clinically significant medical condition.
* Current alcohol/drug use disorder of moderate or severe severity (i.e., subject is not in full remission from moderate to severe alcohol/drug use).
* Two weeks free of antipsychotic medication. (Note: Because a large number of individuals with aggressive tendencies in the community are already taking SSRIs, SNRIs, or mood stabilizers, these individuals will not be excluded if they continue to report impulsive aggressive behaviors at time of study.)
* Unwilling/unable to sign informed consent document.

Ages: 21 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2022-09-06 (Actual); Primary Completion 2027-08-31 (Estimated); Study Completion 2027-08-31 (Estimated)

PRIMARY OUTCOMES:
Cortico-Limbic Response to Anger Faces | 24 hours after Nitrous Oxide and Room Air
  Orbito-Frontal and Amygdala responses to Anger Faces in fMRI
Brain Connectivity | 24 hours after Nitrous Oxide and Room Air
  Resting State

CONTACTS AND LOCATIONS:
Overall Officials: Emil Coccaro, M.D., Principal Investigator — Ohio State University
Locations (1):
- Ohio State University Wexner Medical Center, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No